CLINICAL TRIAL: NCT06512493
Title: South East (Zuid Oost) Netherlands Heart Registry (ZON-HR)
Brief Title: South East (Zuid Oost) Netherlands Heart Registry
Acronym: ZON-HR
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Maastricht Universitair Medisch Centrum (Unknown); Zuyderland Medisch Centrum (Other); VieCuri Medical Centre (Other)
Responsible Party: Sponsor
Other Study IDs: METCZ20200185
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Chronic Coronary Syndrome
Keywords: percutaneous coronary intervention; secondary prevention; chronic coronary syndrome; acute coronary syndrome; personalized medicine
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Patients undergoing percutaneous coronary intervention (PCI) for chronic coronary syndrome (CCS) or acute coronary syndrome (ACS) have a residual risk of ischemic events after PCI due to the progression of atherosclerosis in and outside the stented segments. The residual risk is affected by thrombotic, lipid, inflammation and diabetic risk factors. Secondary prevention after PCI is therefore of major importance to reduce complications and improve the patients' prognosis.

Objective: To provide an extensive overview on the quality of secondary prevention and personalized medicine, a consortium in the South East Netherlands has created a PCI registry, the "Zuid Oost Nederland Hart Registratie" (ZON-HR).

DETAILED DESCRIPTION:
Rationale: Patients undergoing percutaneous coronary intervention (PCI) for chronic coronary syndrome (CCS) or acute coronary syndrome (ACS) have a residual risk of ischemic events after PCI due to the progression of atherosclerosis in and outside the stented segments. The residual risk is affected by thrombotic, lipid, inflammation and diabetic risk factors. Secondary prevention after PCI is therefore of major importance to reduce complications and improve the patients' prognosis. Antithrombotic treatment plays a major role in the reduction of thromboembolic events and is therefore key in secondary prevention. However, this treatment increases the risk of bleeding complications. Therefore, a personalized antiplatelet strategy is recommended by the guidelines. Together with the antithrombotic treatment, lipid management is the cornerstone of secondary prevention. As low density lipoproteins cholesterol (LDL-C) increases the risk for atherosclerotic cardiovascular disease, the current ESC guidelines recommend a LDL-C value <1.4mmol/L in patients undergoing PCI. Personalized medicine in which the treatment and lifestyle advice after PCI is adjusted on the patients' risk factors such as high bleeding- or thromboembolic risk, high LDL cholesterol levels, hypertension or the presence of diabetes mellitus (DM) is of major importance to lower the residual risk of complications and revascularisation. However, due to the large amount of risk factors that should be considered, personalized medicine is challenging which can lead to under treatment.

Objective: To maintain and improve quality of care throughout the Netherlands, all interventional centres deliver data regarding patient- and procedural characteristics and follow-up after PCI to the Netherland Heart Registry (NHR). The NHR processes the data and provides these centres with feedback. (16) However, the registration of baseline-, procedural- and follow-up parameters by the NHR is concise and mainly focuses on mortality and (ischemia driven) revascularisation. To enhance the potency of this PCI registry, a consortium in the South East region of the Netherlands has created an extended version: The "Zuid Oost Nederland Hart Registratie" (ZON-HR). With this comprehensive registry, the ZON-HR provides a more extensive overview on the quality of secondary prevention and personalized medicine. Furthermore, the ZON-HR consortium aims to improve secondary prevention post-PCI by stimulating a personalized approach. Also, it will provide a platform for research regarding secondary prevention.

ELIGIBILITY:
No in- or exclusion criteria are applied to gain 100% registration in order to prevent bias.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing PCI are included in the registry. In line with the NHR, failed PCI attempts are considered as a performed PCI as long as a coronary wire has been inserted in the target vessel.
Sampling Method: Probability Sample
Enrollment: 99999 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2050-01-01 (Estimated); Study Completion 2050-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with | 1 or 2 years
  * all- cause mortality
  * Myocardial infarction
  * Stent thrombosis
  * Stroke
  * Revascularisation
  * All bleeding events requiring medical evaluation

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - ZuyderlandMC, Heerlen, Limburg
  - MaastrichtUMC+, Maastricht, Limburg
  - VieCuri, Venlo, Limburg
  - Radboud University Medical Centre, Nijmegen